CLINICAL TRIAL: NCT02849275
Title: The Effects of Probiotics on Behavioral and Biological Markers of Cognition and Stress
Brief Title: Effects of Probiotics on Cognition and Health
Acronym: EPOCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Hannah Holscher, Assistant Professor of Nutrition, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16840-1
Record Dates: First submitted 2016-07-22; First posted 2016-07-29 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-07

CONDITIONS: Physiological Stress; Cognition - Other
MeSH Terms: interventions — Milk

STUDY DESIGN:
Intervention Model Description: Participants will pass through 2 arms, control and probiotic, in a randomized, counter-balanced order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactose free 1% milk (Placebo Comparator): Diet will be recorded with a 7-day diet record and participants will include an isocaloric study treatment containing lactose free 1% milk consumed once daily over 4-5 weeks as a control.
  Interventions: Other: Lactose Free 1% Milk
- Probiotic treatment (Experimental): Diet will be recorded with a 7-day diet record and participants will include an isocaloric fermented milk (probiotic), consumed once daily, over 4-5 weeks.
  Interventions: Other: Probiotic Treatment

INTERVENTIONS:
Other: Lactose Free 1% Milk — isocaloric study treatment containing lactose free 1% milk consumed once daily over 4-5 weeks as a control.
  Arms: Lactose free 1% milk
Other: Probiotic Treatment — Probiotic treatment, consumed once daily, over 4-5 weeks.
  Arms: Probiotic treatment

SUMMARY:
This research intervention aims to examine the effects of a fermented dairy beverage on changes in behavioral and biological measures of cognition and stress among adults.

DETAILED DESCRIPTION:
Evidence-based dietary strategies provide behavioral means benefiting physical and cognitive function. Pertinent to the proposed work, dietary intake has been recently shown to have the potential to directly influence the gut microbiota composition as well as brain function. Specifically, the consumption of probiotics or foods containing healthful microbial cultures (e.g., fermented milk, yogurts, etc.) are increasingly being recognized as modulators of metabolism, cognition, and stress. These foods are readily available in the marketplace, however, their implications for physical and cognitive function are not clear. Accordingly, the proposed study aims to investigate effects of probiotic beverage consumption on changes in behavioral and biological measures of cognition and stress among adults.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Between the ages of 25-45 years at the time of consent
* BMI ≥18.5 kg/m2
* Normal or corrected-to-normal vision based on the minimal 20/20 standard in order to complete the cognitive task.
* Ability to drop-off fecal sample within 15 minutes of defecation

Exclusion Criteria:

* Current pregnancy or lactation
* Tobacco use
* Dairy allergy or intolerance
* Prior diagnosis of metabolic and gastrointestinal disease (cardiovascular disease and type 1 or type 2 diabetes, chronic constipation, diarrhea, Crohn's disease, celiac disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis, HIV, cancer, etc.)
* Prior diagnosis of cognitive or physical disability, including ADHD, severe asthma, epilepsy, chronic kidney disease
* Use of any anti-psychotic, anti-depressant, anti-anxiety, or ADD/ADHD medications
* Use of medications that alter normal bowel function and metabolism (e.g., recent antibiotic use, laxatives, enemas, anti-diarrheal agents, narcotics, antacids, antispasmodics, diuretics, anticonvulsants).
* Prior malabsorptive bariatric surgery (i.e. gastric bypass, sleeve gastrectomy) or restrictive bariatric surgery (i.e. adjustable gastric band) within the past 2 years.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Changes in cortisol as a biomarker of stress | 4-5 weeks
  The effects of probiotic consumption on biomarkers of stress

SECONDARY OUTCOMES:
Changes in fecal microbiota populations | 4-5 weeks
  The effects of probiotic consumption on fecal microbiota

OTHER OUTCOMES:
Changes in cognition | 4-5 weeks
  The effects of probioticconsumption on cognition

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Holscher, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign; Naiman Khan, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be disseminated by journal articles, thesis or academic papers, conference presentations, and sharing with the funding organization. No subject's identity will be disclosed in any presentation or released without their written permission.

REFERENCES:
- [Derived] Cannavale CN, Mysonhimer AR, Bailey MA, Cohen NJ, Holscher HD, Khan NA. Consumption of a fermented dairy beverage improves hippocampal-dependent relational memory in a randomized, controlled cross-over trial. Nutr Neurosci. 2023 Mar;26(3):265-274. doi: 10.1080/1028415X.2022.2046963. Epub 2022 Mar 13. PMID 35282787